CLINICAL TRIAL: NCT06176937
Title: Efficacy of Hyaluronic Acid Gel in Ridge Preservation After Tooth Extraction: A Randomized Controlled Clinical Trial With Radiographic and Histomorphometric Study
Brief Title: Hyaluronic Acid Gel in Ridge Preservation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FD-ASU-REC.852
Record Dates: First submitted 2023-09-13; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2020-01

CONDITIONS: Hyaluronic Acid Gel for Preservation the Extraction Socket
Keywords: hopeless anterior tooth; atraumatic extraction; hyaluronic acid gel
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyaluronic acid gel (Active Comparator): Hyaluronic acid considers as a high molecular weight glycosaminoglycan (GAG) consists of multiple disaccharide non-sulfated units of D-glucuronic acid and N-acetylglucosamine
  Interventions: Drug: Hyaluronic acid
- empty socket (Other): extraction socket without application any drug
  Interventions: Other: empty socket

INTERVENTIONS:
Drug: Hyaluronic acid — Alveolar ridge preservation by atraumatic tooth extraction and socket curettage then application hyaluronic acid gel after extraction and covering the socket by collagen membrane.
  Arms: hyaluronic acid gel
Other: empty socket — Alveolar ridge preservation by atraumatic tooth socket without application any drug but just covering the socket by collagen membrane.
  Arms: empty socket

SUMMARY:
hyaluronic acid gel applied at the extraction socket after extraction immediately to preserve the socket from post extraction resorption. hyaluronic acid has ability for osteogenesis and new bone formation.

DETAILED DESCRIPTION:
twenty-four patients with one hopeless tooth at least, first CBCt before extraction to evaluate the dimension of the socket, then atraumatic extraction of the tooth to preserve the bony wall of the socket, after extraction and curettage the socket applied hyaluronic acid gel inside the socket and applied collagen membrane to secure the socket. After 4 months of extraction, CBCt was done to evaluate the dimension of the socket and the effect of hyaluronic acid. Furthermore, The core biopsy was taken by trephine bur at the time of implant placement for evaluate the histological appearance of the bone to evaluate the secondary outcome. then after three months the crown was delivered as a prosthetic part.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult patients as evidenced by Burkett's oral medicine health history questionnaire
2. Both genders.
3. Age from 20 -50 years old.
4. Having at least one hopeless teeth indicated for extraction.
5. Esthetic zone teeth (anterior or premolar).
6. Sockets type 1 or 2 .
7. Patient should agree to sign a written consent after the nature of the study will be explained.

   -

   Exclusion Criteria:

1- Smokers. 2- Pregnant and breast-feeding females. 3- Mentally retarded Patients. 4- Prisoners and handicapped patients. 5- Patients with malocclusion.

-

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
clinical outcome | baseline(before extraction)/ four months later after extraction
  measurement clinical bone width of the socket by millimeter before and 4 months after extraction ...
Radiographic measurement | baseline(before extraction)/ four months later after extraction
  Radiographic measurement of bone width by CBCt before and 4 months after extraction
Radiographic measurement | baseline (before extraction)/ four months later after extraction
  Radiographic measurement of bone height by CBCt before and 4 months after extraction.

SECONDARY OUTCOMES:
histological analysis | after 4 months of extraction at the time of implant placement.
  The bone biopsy will be taken by trephine bur. And evaluate bone quality.
histomorphometric analysis | after 4 months of extraction at the time of implant placement.
  The bone biopsy will be taken by trephine bur. And evaluate bone quantity.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan M Ibrahim, professor, Study Director — Faculty of dentistry-Ain shams university
Locations (1):
- Ain shams University, Cairo, Egypt